CLINICAL TRIAL: NCT03742518
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of 0.15% & 0.25% Concentrations of Topical SM04554 Solution in Male Subjects With Androgenetic Alopecia
Brief Title: A Study Evaluating the Efficacy and Safety of SM04554 Topical Solution in Male Subjects With Androgenetic Alopecia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SM04554-AGA-05
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Androgenetic Alopecia
Keywords: male pattern baldness; SM04554; AGA
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Topical SM04554 0.15% solution (Experimental): Topical SM04554 0.15% solution, once daily for up to 48 weeks
  Interventions: Drug: Topical SM04554 solution
- Topical SM04554 0.25% solution (Experimental): Topical SM04554 0.25% solution, once daily for up to 48 weeks
  Interventions: Drug: Topical SM04554 solution
- Vehicle (Placebo Comparator): Topical vehicle solution, once daily for up to 48 weeks
  Interventions: Drug: Topical vehicle solution

INTERVENTIONS:
Drug: Topical SM04554 solution — Study medication application will be performed by the individual subject at approximately the same time each day.
  Arms: Topical SM04554 0.15% solution
Drug: Topical SM04554 solution — Study medication application will be performed by the individual subject at approximately the same time each day.
  Arms: Topical SM04554 0.25% solution
Drug: Topical vehicle solution — Vehicle solution application will be performed by the individual subject at approximately the same time each day.
  Arms: Vehicle

SUMMARY:
This multi-center, randomized, double-blind, placebo-controlled study, conducted in Turkey, will assess the efficacy and safety of topical SM04554 solution (0.15% and 0.25%) applied daily to the scalp of male androgenetic alopecia (AGA) subjects.

ELIGIBILITY:
Inclusion Criteria:

* Being a Turkish citizen
* Clinical diagnosis of AGA with Norwood-Hamilton Classification score of 3V or 4
* Willing to inform females, with whom they may interact, that they are using a topical investigational product and direct contact should be avoided as potential harm to a fetus is unknown
* Willing and able to attend all study visits
* Willing to maintain the same hair style and length as at the study start for the duration of the study
* Willing to not use semi-permanent hair products (e.g., color, texturizers, relaxers) for the duration of the study; daily styling products (e.g., hair gel, mousse, styling spray) will be allowed on non-study visit days
* Willing to use mild non-medicated shampoo and conditioner for the duration of the study
* Able to read and understand Turkish
* Ability to comprehend and willing to sign an informed consent form

Exclusion Criteria:

* Males who are sexually active, and have a partner who is capable of becoming pregnant, if neither has had surgery to become sterilized, and/or who are not willing to use condom or whose partner is not using a highly effective method of birth control that includes double barrier, intrauterine device, or hormonal contraceptive combined with single barrier, or abstinence during the study treatment period until 90 days post last dose of study medication
* Clinical diagnosis of alopecia areata or other non-AGA forms of alopecia
* Scalp hair loss on the treatment area, due to disease, injury, or medical therapy
* History of surgical correction (e.g., hair transplantation, scalp reduction) of hair loss on the scalp
* Previous exposure to SM04554
* Use of any products (e.g., finasteride, minoxidil, platelet rich plasma, biotin) or devices (e.g., laser light therapy) purported to promote scalp hair growth within 24 weeks prior to the start of the study
* Use of anti-androgenic therapies (e.g., spironolactone, flutamide, cyproterone acetate, cimetidine) within 12 weeks prior to the start of the study
* Use of medications that potentially cause drug-induced hair loss (e.g., depotestosterone, haloperidol, methotrexate, methylprednisolone, prednisone, testosterone, divalproex sodium) within 12 weeks prior to the start of the study
* Current use of an occlusive wig, hair extensions, or hair weaves
* History of hypersensitivity or allergies to any ingredient of the study medication
* Participation in any other investigational drug or medical device trial, which includes or included administration of an investigational study medication or medical device, within 30 days or 5 half-lives of the investigational agent, whichever is longer, prior to the start of the study
* Use of semi-permanent hair products (e.g., color, texturizers, relaxers) within 30 days prior to the start of the study
* Use of medicated shampoo or conditioner (medicated shampoo and conditioner refers to any prescription shampoo or conditioner as well as any over-the-counter medicated shampoo or conditioner, such as those for treatment of dandruff or promoting hair growth) within 30 days prior to the start of the study
* Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the investigative site, or are directly affiliated with the study at the investigative site
* Subjects employed by Samumed, LLC or Samumed Turkey, or any of its affiliates or development partners (i.e., an employee, temporary contract worker, or designee) responsible for the conduct of the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 675 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Absolute non-vellus hair count in target area | Week 48
  Absolute non-vellus hair count in target area by phototrichogram (PTG) analysis

SECONDARY OUTCOMES:
Absolute non-vellus hair count in target area | Weeks 12, 24, and 36
  Absolute non-vellus hair count in target area by PTG analysis
Absolute vellus hair count in target area | Weeks 12, 24, 36 and 48
  Absolute vellus hair count in target area by PTG analysis
Absolute total hair count in target area | Weeks 12, 24, 36 and 48
  Absolute total hair count in target area by PTG analysis
Change from baseline in non-vellus hair count in target area | Baseline, and Weeks 12, 24, 36 and 48
  Change from baseline in non-vellus hair count in target area by PTG analysis
Change from baseline in vellus hair count in target area | Baseline, and Weeks 12, 24, 36 and 48
  Change from baseline in vellus hair count in target area by PTG analysis
Change from baseline in total hair count in target area | Baseline, and Weeks 12, 24, 36 and 48
  Change from baseline in total hair count in target area by PTG analysis
Change from baseline in average non-vellus hair shaft thickness in target area | Baseline, and Weeks 12, 24, 36 and 48
  Change from baseline in average non-vellus hair shaft thickness in target area by PTG analysis
Change from baseline in average non-vellus hair density in target area | Baseline, and Weeks 12, 24, 36 and 48
  Change from baseline in average non-vellus hair density (cumulative non-vellus hair shaft thickness) in target area by PTG analysis
Subject assessment of hair growth | Weeks 6, 12, 18, 24, 30, 36, 42 and 48
  Subjects will complete a questionnaire for hair growth while referencing the global scalp photograph taken at the visit as compared to their baseline global scalp photograph. The scale for the questionnaire ranges from -3 to +3 (-3 indicates the worst outcome and +3 indicates the best outcome).
Change from baseline in subject assessment of hair satisfaction | Baseline, and Weeks 6, 12, 18, 24, 30, 36, 42 and 48
  Subjects will complete a questionnaire for hair satisfaction while referencing the global scalp photograph taken at the visit as compared to their baseline global scalp photograph. The scale for the questionnaire ranges from -3 to +3 (-3 indicates the worst outcome and +3 indicates the best outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (11):
- Turkey (Türkiye) (11):
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Denizli
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kayseri
  - Research Site, Kocaeli
  - Research Site, Mersin
  - Research Site, Samsun
  - Research Site 1, Trabzon
  - Research Site 2, Trabzon